CLINICAL TRIAL: NCT03948828
Title: Clinical Study on the Treatment of Endometriosis by Combining With the Pathogenesis of Endometriosis and the Application Characteristics of NK Cells
Brief Title: Clinical Study of NK Cells in the Treatment of Severe Endometriosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShenzhenPH BTR-003
Record Dates: First submitted 2019-03-28; First posted 2019-05-14 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: NK Cell Mediated Immunity; Endometriosis
Keywords: Endometriosis; NK cell therapy
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment group (Other): GnRHa combained with reverse addition therapy
  Interventions: Drug: GnRHa combained with reverse addition therapy
- Conventional treatment and Autologous NK cells therapy (Experimental): GnRHa combained with reverse addition therapy and NK cell combined treatment group
  Interventions: Biological: Autologous NK cell therapy; Drug: GnRHa combained with reverse addition therapy

INTERVENTIONS:
Biological: Autologous NK cell therapy — After conventional treatment, the patients were treated with autologous NK cells.
  Arms: Conventional treatment and Autologous NK cells therapy
Drug: GnRHa combained with reverse addition therapy — Postoperative patients were treated with GnRHa combined with reverse addition treatment.
  Other Names: Conventional treatment

SUMMARY:
Dysfunction of natural koller cells (NK cells) is an important factor in the development of endometriosis. NK cell therapy was applied to treat severe endometriosis, which is an exploration of the pathogenesis of this refractory disease.

DETAILED DESCRIPTION:
Endometriosis (EMs) is one of the common and frequently occurring diseases in women of childbearing age, which seriously affects the health and quality of life of the vast majority of women. The pathogenesis of endometriosis is unknown until now, and the recurrence rate of existing treatment methods is high. It is more and more necessary to introduce new therapeutic methods and strategies in view of the mechanism associated with the reduction of natural killer cell (NK) cytotoxicity. In this study, routine therapy combined with NK cell therapy was used in the treatment of severe endometriosis. The clinical data were collected to confirm the efficacy and safety of NK cell therapy. It is expected to provide a new way of thinking and method for the clinical treatment of EMs.

ELIGIBILITY:
Inclusion Criteria:

1. Diagonsed as endometriosis stage III~IV
2. Age ≥18 years ≤ 45 years at the time of informed consent
3. With indications for conservative endometriosis surgery
4. With complete clinical data

Exclusion Criteria:

1. Severe allergy to drugs
2. Patients with abnormal immune status (Autoimmune disease or long-term use of immunosuppressive agents)
3. With serious cardiac, cerebrovascular diseases and liver, kidney disorders
4. With a history of severe mental illness

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety] | 3 months after treatment
  Adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events v4.0
Purity and Function of NK cells | once per three months
  The purity and function of NK cells will be measured by flow cytometry.

SECONDARY OUTCOMES:
Endocrine hormone levels | every three months, up to 36 months
  The levels of endocrine hormone, including serum estradiol, testosterone, progesterone, luteinizing hormone and follicle stimulating hormone will be measured.
Pain score | every three months, up to 36 months
  A score of 0 means that you have never had this problem, and a score of 100 means that you are always troubled by this problem and feel unbearable. You can choose any number between 0 and 100 to represent your feelings. The higher the score, the worse your feelings will be.
The percent of pregnancy | 36 months
  The pregnancy will be meaured by B ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Qi, M.D, Study Director — Shen Zhen People's Hospital
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No